CLINICAL TRIAL: NCT04094272
Title: Pulmonary Arterial Hypertension in Patients With Direct-Acting Antiviral Medications for Hepatitis C Virus Infection - a Prospective Observational Cohort Study
Brief Title: Pulmonary Arterial Hypertension in Patients With Direct-Acting Antiviral Medications for Hepatitis C Virus Infection
Status: Completed | Type: Observational
Sponsor: Kantonsspital Olten (Other)
Responsible Party: Principal Investigator, Nisha Arenja, Head of Cardiovascular Imaging, Kantonsspital Olten
Other Study IDs: PAH-HCV
Record Dates: First submitted 2019-09-16; First posted 2019-09-18 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Pulmonary Artery Hypertension; Chronic Hepatitis c
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension; Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic hepatitis C participants: Participants with a newly started DAA medication for HCV infection were included in the study.
  Interventions: Diagnostic Test: transthoracic doppler-echocardiography (TTE)

INTERVENTIONS:
Diagnostic Test: transthoracic doppler-echocardiography (TTE) — Transthoracic doppler-echocardiography (TTE) in patients with a new diagnosis of HCV before and after treatment with DAA medication.

SUMMARY:
The purpose of this study is the evaluation of PAH in patients, who are treated with DAA medication for HCV infection.

DETAILED DESCRIPTION:
Study category and Rationale: This study is without any use of medication or investigations products, therefore this is a category A clinical trail.

Background and Rationale: Pulmonary arterial hypertension (PAH) is a chronic and progressive disease leading to right heart failure and ultimately death in untreated patients. A variety of systemic illnesses have been associated with PAH. Hepatitis C virus (HCV) infection is not defined as a risk factor for PAH. However, compared to a control population higher pulmonary artery pressures are described in patients with HCV. Some case reports indicate association between HCV medication and PAH. Except of a few case reports, to date no clinical study about evidence of PAH in patients with direct-acting-antiviral (DAA) medication for HCV infection has been published.

Objective: The purpose of this study is the evaluation of PAH in patients, who are treated with DAA medication for HCV infection.

Outcomes: The primary outcome of this study is the evaluation of pulmonary artery pressure change using transthoracic doppler-echocardiography (TTE) in patients with a new diagnosis of HCV before and after treatment with DAA medication. The secondary outcomes are the change in left and right ventricular structure and function using TTE in patients with a new diagnosis of HCV before and after treatment with DAA medication.

Study design: A single center prospective, observational cohort study. Inclusion / Exclusion criteria: Inclusion criteria are evidence of HCV infection and age 18-90 years. Patients will be excluded from the study, if there is an inability to provide informed consent and if there are known for existing PAH.

Measurements and procedures: The patients will receive a TTE for the measurement of the pulmonary artery pressure before, during (8 weeks after starting the medication) and 8 weeks after completion of the HCV medication. The whole treatment period will take about 12 weeks.

Study Product / Intervention: The study will use a TTE for measurement of pulmonary artery pressure. This non-invasive, fast investigation (total duration about 20 minutes) is used for years in Cardiology and does not constitute a specific study product.

Number of Participants with Rationale:The study goal ist the înlusion of 50 participants with a newly started DAA medication for HCV infection. Due to the lack of data, a power calculation is not possible. However, if a higher number than 50 participants would be necessary to show a significant rise in pulmonary pressure, a clinical significance is not likely to be relevant.

Study Duration: The study inclusion is planned for 2 year.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-90 years
* Written informed consent
* New diagnosis of HCV, which requires the initiation of a DAA therapy

Exclusion Criteria:

* Inability to provide informed consent
* Known diagnosis of pulmonary artery hypertension (PAH)
* Dyspnoe NYHA III-IV
* Mean pulmonary artery (PA) pressure (mPAP) of >25 mmHg in the first TTE before start of DAA medication

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — self-representation of gender identity
Study Population: All patients who will assign or present with diagnosis of HCV to the infectologist at the Kantonsspital Olten, (community clinic) wasl asked to take part in the study.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Assessment of pulmonary artery pressure | 2 years
  evaluation of pulmonary artery pressure change using transthoracic doppler-echocardiography (TTE

SECONDARY OUTCOMES:
Left and right ventricular structure and function | 2. years
  The secondary outcomes are the change in left and right ventricular structure and function using TTE in patients with a new diagnosis of HCV before and after treatment with DAA medication.

CONTACTS AND LOCATIONS:
Locations (1):
- Kantonsspital Olten, Olten, Switzerland

IPD SHARING:
Plan to Share IPD: No